CLINICAL TRIAL: NCT03097133
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Intranasal Esketamine in Addition to Comprehensive Standard of Care for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation, in Adult Subjects Assessed to be at Imminent Risk for Suicide
Brief Title: 54135419SUI3002: A Study to Evaluate the Efficacy and Safety of Intranasal Esketamine in Addition to Comprehensive Standard of Care for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation, in Adult Participants Assessed to be at Imminent Risk for Suicide
Acronym: Aspire II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108285; 2016-003992-23 (EudraCT Number); 54135419SUI3002 (Other: Janssen Research & Development, LLC)
Expanded Access: NCT03829579 (Approved for marketing)
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Esketamine; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Esketamine + Standard of care (Experimental): Participants will receive intranasal esketamine 84 milligram (mg) on Day 1, 4, 8, 11, 15, 18, 22, and 25 along with standard of care antidepressant treatment.
  Interventions: Drug: Esketamine; Other: Standard of Care
- Placebo + Standard of care (Placebo Comparator): Participants will receive intranasal placebo on Day 1, 4, 8, 11, 15, 18, 22, and 25 along with standard of care antidepressant treatment.
  Interventions: Drug: Placebo; Other: Standard of Care

INTERVENTIONS:
Drug: Esketamine — Participants will receive intranasal esketamine 84 milligram (mg) two times per week for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25).
  Arms: Esketamine + Standard of care
Drug: Placebo — Participants will receive intranasal placebo two times per week for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25).
  Arms: Placebo + Standard of care
Other: Standard of Care — The standard of care antidepressant treatment (antidepressant monotherapy or antidepressant plus augmentation therapy) will be determined by the treating physician(s) based on clinical judgement and practice guidelines prior to randomization, and the treatment will be initiated on Day 1.

SUMMARY:
The purpose of this study is to evaluate the efficacy of intranasal esketamine 84 milligram (mg) compared with intranasal placebo in addition to comprehensive standard of care in reducing the symptoms of Major Depressive Disorder (MDD), including suicidal ideation, in participants who are assessed to be at imminent risk for suicide, as measured by the change from baseline on the Montgomery-Asberg Depression Rating Scale (MADRS) total score at 24 hours post first dose.

DETAILED DESCRIPTION:
If you or a loved one are having thoughts of suicide, please seek immediate medical help. Go to the emergency room or call the National Suicide Prevention Lifeline at 1-800-273-8255.

ELIGIBILITY:
Inclusion Criteria:

* Participant must meet Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) diagnostic criteria for major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the Mini International Psychiatric Interview (MINI)
* Participants must have current suicidal ideation with intent, confirmed by a "Yes" response to Question B3 [Think (even momentarily) about harming or of hurting or of injuring yourself: with at least some intent or awareness that you might die as a result; or think about suicide (ie, about killing yourself)?] AND Question B10 [Intend to act on thoughts of killing yourself?] obtained from the MINI
* In the physician's opinion, acute psychiatric hospitalization is clinically warranted due to participant's imminent risk of suicide
* Participant has a Montgomery Asberg Depression Rating Scale (MADRS) total score of greater than (>) 28 predose on Day 1
* As part of standard of care treatment, participant agrees to be hospitalized voluntarily for a recommended period of 14 days after randomization (may be shorter or longer if clinically warranted in the investigator's opinion) and take prescribed non-investigational antidepressant therapy(ies) for at least the duration of the double-blind treatment phase (Day 25)

Exclusion Criteria:

* Participant has a current DSM-5 diagnosis of bipolar (or related disorders), antisocial personality disorder, or obsessive compulsive disorder
* Participant currently meets DSM-5 criteria for borderline personality disorder. Note: Participant not meeting full DSM-5 criteria for borderline personality disorder but exhibiting recurrent suicidal gestures, threats, or self-mutilating behaviors should also be excluded
* Participant has a current clinical diagnosis of autism, dementia, or intellectual disability
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder, or MDD with psychotic features
* Participant meets the DSM-5 severity criteria for moderate or severe substance or alcohol use disorder, (except for nicotine or caffeine), within the 12 months before Screening. A history (lifetime) of ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3, 4-methylenedioxy-methamphetamine (MDMA) hallucinogen-related use disorder is exclusionary
* Participant has a history or current signs and symptoms of liver or renal insufficiency, clinically significant cardiac (including unstable coronary artery disease and congestive heart failure, tachyarrhythmias and recent myocardial infarction) or vascular, pulmonary, gastrointestinal, endocrine (including uncontrolled hyperthyroidism), neurologic (including current or past history of seizures except uncomplicated childhood febrile seizures with no sequelae), hematologic, rheumatologic, or metabolic (including severe dehydration/ hypovolemia) disease
* Participant has known allergies, hypersensitivity, intolerance or contraindications to esketamine or ketamine or its excipients

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (61):
- United States (18):
  - University of California San Diego/Psychiatry, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - University of Conneticut School of Medicine, Farmington, Connecticut
  - University of Miami Health System, Miami, Florida
  - Innovative Clinical Research Inc, North Miami, Florida
  - University of South Florida, Tampa, Florida
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - Memorial Medical Center, Springfield, Illinois
  - Neuroscience Research Institute, Winfield, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - John Hopkins Hospital, Baltimore, Maryland
  - Altea Research Institute, Las Vegas, Nevada
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Cincinnati, Dept of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio
  - East Tennessee State University, Johnson City, Tennessee
  - University of Wisconsin Medical Center, Madison, Wisconsin
- Argentina (4):
  - Clínica Privada Banfield S.A, Banfield
  - Hospital Fleni, Ciudad de Buenos Aires
  - Sanatorio Prof. Leon S. Morra, Córdoba
  - Clinica Privada de Salud Mental Santa Teresa de Ávila, La Plata
- Austria (2):
  - Medical University Vienna MUV, Vienna
  - Klinikum Wels Grieskirchen, Wels
- Belgium (3):
  - AZ Sint Jan Brugge Oostende AV, Bruges
  - UZ Gent, Ghent
  - ARIADNE, Lede
- Brazil (6):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Universidade Federal Do Ceara, Fortaleza
  - Instituto Bairral de Psiquiatria, Itapira
  - Hospital Universitario Professor Edgar Santos, Salvador
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, Santo André
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Institut universitaire en sante mentale de Montreal, Montreal, Quebec
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Nemocnice s pol. Havirov, p.o., Havířov
  - Narodni ustav dusevniho zdravi, Klecany
  - Vseobecna Fakultní Nemocnice, Prague
  - Ústrední vojenské nemocnice Praha, Prague
- France (6):
  - Hôpital de Bohars, Bohars
  - CHRU Montpellier Hopital Lapeyronie, Montpellier
  - CHU Caremeau, Nîmes
  - Hopital Sainte Anne, Paris
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHU Toulouse, Toulouse
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Republic Kaunas Hospital, Kaunas County
  - Vilnius Mental Health Center, Vilnius
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Specjalistyczny im H Klimontowicza Oddzial Psychiatryczny, Gorlice
  - SPZOZ CSK UM w Lodzi Klinika Zaburzen Afektywnych i Psychotycznych, Lodz
  - Klinika Psychiatryczna WUM Mazowieckie Specjalistyczne Centrum Zdrowia im prof Jana Mazurkiewicza, Pruszków
- Spain (4):
  - Hosp Univ Vall D Hebron, Barcelona
  - Inst. Internac. Neurociencias Aplicadas, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Clinica Univ. de Navarra, Pamplona
- Turkey (Türkiye) (4):
  - Bursa Sevket Yilmaz Research and Training Hospital, Bursa
  - Uludag University Medical Faculty, Bursa
  - Sisli Etfal Research Training Hospital, Istanbul
  - Samsun Psychiatric Hospital, Samsun

REFERENCES:
- [Derived] Fu DJ, Zhang Q, Shi L, Borentain S, Guo S, Mathews M, Anjo J, Nash AI, O'Hara M, Canuso CM. Esketamine versus placebo on time to remission in major depressive disorder with acute suicidality. BMC Psychiatry. 2023 Aug 11;23(1):587. doi: 10.1186/s12888-023-05017-y. PMID 37568081
- [Derived] Jamieson C, Canuso CM, Ionescu DF, Lane R, Qiu X, Rozjabek H, Molero P, Fu DJ. Effects of esketamine on patient-reported outcomes in major depressive disorder with active suicidal ideation and intent: a pooled analysis of two randomized phase 3 trials (ASPIRE I and ASPIRE II). Qual Life Res. 2023 Nov;32(11):3053-3061. doi: 10.1007/s11136-023-03451-9. Epub 2023 Jul 13. PMID 37439961
- [Derived] Turkoz I, Lopena O, Salvadore G, Sanacora G, Shelton R, Fu DJ. Treatment response to esketamine nasal spray in patients with major depressive disorder and acute suicidal ideation or behavior without evidence of early response: a pooled post hoc analysis of ASPIRE. CNS Spectr. 2023 Aug;28(4):482-488. doi: 10.1017/S1092852922000931. Epub 2022 Jul 29. PMID 35904046
- [Derived] Rozjabek H, Li N, Hartmann H, Fu DJ, Canuso C, Jamieson C. Assessing the meaningful change threshold of Quality of Life in Depression Scale using data from two phase 3 studies of esketamine nasal spray. J Patient Rep Outcomes. 2022 Jul 10;6(1):74. doi: 10.1186/s41687-022-00453-y. PMID 35816217
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Ionescu DF, Fu DJ, Qiu X, Lane R, Lim P, Kasper S, Hough D, Drevets WC, Manji H, Canuso CM. Esketamine Nasal Spray for Rapid Reduction of Depressive Symptoms in Patients With Major Depressive Disorder Who Have Active Suicide Ideation With Intent: Results of a Phase 3, Double-Blind, Randomized Study (ASPIRE II). Int J Neuropsychopharmacol. 2021 Jan 20;24(1):22-31. doi: 10.1093/ijnp/pyaa068. PMID 32861217
- See also: A Study to Evaluate the Efficacy and Safety of Intranasal Esketamine in Addition to Comprehensive Standard of Care for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation (Aspire II) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108285&attachmentIdentifier=6345e95c-007a-4ab5-b5f6-736c8099e66f&fileName=54135419SUI3002_(CR108285)_Additional_Results_Data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Standard of Care (SOC): Participants self-administered intranasal placebo (1 spray in each nostril at 0, 5 and 10 minutes using 3 devices on a single day) twice per week for 4 weeks on days 1, 4, 8, 11, 15, 18, 22, and 25 along with SOC antidepressant treatment (determined by the physician based on clinical judgment and practice guidelines) on Day 1 and continued for the duration of the double-blind (DB) treatment phase (Days 1 to 25).
- Esketamine 84 mg + SOC: Participants self-administered esketamine 84 milligram (mg) (1 spray containing esketamine 14 mg in each nostril at 0, 5, 10 minutes using 3 devices on single day) twice per week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, 25 along with SOC antidepressant treatment (determined by physician based on clinical judgment and practice guidelines) on Day 1 continued for DB treatment phase. After Day 1, a single dose reduction from esketamine 84 mg to 56 mg was permitted if a participant was unable to tolerate intranasal esketamine 84 mg dose. Participants for whom dose was reduced continued to receive reduced dose for duration of DB treatment phase (Days 1 to 25).
Period: Overall Study
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Started | 115 | 115
Treated | 113 | 114
Completed | 85 | 81
Not Completed | 30 | 34
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Discontinued DB, not entered FU Phase | 21 | 25
Not completed — Other | 3 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full efficacy analysis set included all randomized participants who received at least 1 dose of intranasal study agent during DB treatment phase and had both baseline and post baseline evaluation for Montgomery-Asberg Depression Rating Scale (MADRS) total score or Clinical Global Impression - Severity of Suicidality - Revised (CGI-SS-R).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC | Total
Number analyzed (Participants) | 113 | 114 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (13.43) | 40.2 (12.73) | 40.8 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 69 | 136
  Male | 46 | 45 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 7 | 15
  White | 87 | 92 | 179
  More than one race | 6 | 8 | 14
  Unknown or Not Reported | 8 | 6 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 9 | 7 | 16
  AUSTRIA | 5 | 4 | 9
  BELGIUM | 2 | 1 | 3
  BRAZIL | 18 | 18 | 36
  CANADA | 1 | 0 | 1
  CZECH REPUBLIC | 2 | 1 | 3
  FRANCE | 9 | 15 | 24
  LITHUANIA | 1 | 2 | 3
  POLAND | 15 | 18 | 33
  SPAIN | 5 | 5 | 10
  TURKEY | 10 | 13 | 23
  UNITED STATES | 36 | 30 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at 24 Hours Post First Dose (Last Observation Carried Forward [LOCF] Data): Double-blind (DB) Treatment Phase
Description: MADRS is clinician-rated scale designed to be used in participants with Major Depressive Disorder (MDD) to measure depression severity and detect changes due to antidepressant treatment. It evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic and suicidal thoughts. Scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms), summed for total possible score of 0 to 60. Higher scores represent more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1, predose) and 24 hours first post dose (Day 2)
Population: Full efficacy analysis set included all randomized participants who received at least 1 dose of intranasal study agent during DB treatment phase and had both baseline and post baseline evaluation for MADRS total score or CGI-SS-R. Here, 'N' (number of participants analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 113
units on a scale | -12.4 (10.43) | -15.7 (11.56)
Statistical Analysis 1: Comparison: Placebo + Standard of Care (SOC) vs Esketamine 84 mg + SOC; Test type: Superiority; p = 0.006, ANCOVA; Difference of Least Square Means = -3.9, 95% CI 2-sided [-6.60 to -1.11], Standard Error of Mean 1.39

2. Primary Outcome: Change From Baseline in Clinical Global Impression-Severity of Suicidality - Revised (CGI-SS-R) Scale at 24 Hours Post First Dose (LOCF Data): DB Treatment Phase
Description: Clinical global impression-severity of suicidality-revised (CGI-SS-R) scale is revised version of the clinical global impression severity scale (CGI-S),a global rating scale that gives an overall measure of the severity of a participants illness. The CGI-SS-R summarizes the clinician's overall impression of severity of suicidality on a 7-point scale from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal participants), based on the totality of information available to the clinician. Higher score indicates a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1, predose) and 24 hours first post dose (Day 2)
Population: Analysis was performed on full efficacy analysis set. Here 'N' (number of participants analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 113
units on a scale | -1.0 [-5 to 2] | -1.0 [-6 to 2]

3. Secondary Outcome: Number of Participants With Remission of Major Depressive Disorder (MADRS Total Score Less Than or Equal to [<=] 12): DB Treatment Phase
Description: as for outcome 1
Time Frame: Days 1 (4 hours [h] postdose), 2, 4, 8, 11, 15, 18, 22 and 25 (predose and 4 hours postdose)
Population: Analysis was performed on full efficacy analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
Participants
  Day 1: 4 hours post dose | 4 | 12
  Day 2 | 12 | 25
  Day 4 | 20 | 26
  Day 8 | 23 | 28
  Day 11 | 26 | 32
  Day 15 | 29 | 36
  Day 18 | 32 | 29
  Day 22 | 37 | 42
  Day 25: Predose | 31 | 49
  Day 25: 4 hours postdose | 42 | 54

4. Secondary Outcome: Change From Baseline in MADRS Total Score at 4 Hours Post First Dose at Day 1 (4 Hours Post First Dose), and 2, 4, 8, 11, 15, 18, 22 and 25: DB Treatment Phase
Description: MADRS is a clinician-rated scale designed to be used in participants with MDD to measure depression severity and detect changes due to antidepressant treatment. MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts. The instrument consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 0 to 60. Higher scores represent a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1, predose), Days 1 (4 hours postdose), 2, 4, 8, 11, 15, 18, 22 and 25 (predose and 4 hours postdose)
Population: Analysis was performed on full efficacy analysis set. Here 'n' (number analyzed) signifies number of participants analyzed for each specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 1: 4 hours postdose: number analyzed (Participants) | 112 | 112
  Change at Day 1: 4 hours postdose | -8.2 (7.62) | -12.2 (9.87)
  Change at Day 2: number analyzed (Participants) | 111 | 110
  Change at Day 2 | -12.4 (10.51) | -16.0 (11.52)
  Change at Day 4: number analyzed (Participants) | 111 | 107
  Change at Day 4 | -15.7 (11.50) | -17.7 (11.94)
  Change at Day 8: number analyzed (Participants) | 105 | 99
  Change at Day 8 | -17.4 (11.29) | -20.1 (11.47)
  Change at Day 11: number analyzed (Participants) | 99 | 95
  Change at Day 11 | -19.5 (11.60) | -21.3 (11.45)
  Change at Day 15: number analyzed (Participants) | 99 | 91
  Change at Day 15 | -20.0 (12.54) | -23.4 (10.62)
  Change at Day 18: number analyzed (Participants) | 90 | 84
  Change at Day 18 | -21.4 (12.90) | -23.1 (11.39)
  Change at Day 22: number analyzed (Participants) | 94 | 90
  Change at Day 22 | -22.0 (12.12) | -24.5 (11.57)
  Change at Day 25: Predose: number analyzed (Participants) | 88 | 85
  Change at Day 25: Predose | -22.5 (12.23) | -26.2 (11.09)
  Change at Day 25: 4 hours postdose: number analyzed (Participants) | 87 | 83
  Change at Day 25: 4 hours postdose | -26.4 (11.18) | -28.7 (10.88)

5. Secondary Outcome: Change From Baseline in CGI-SS-R Score at 4 Hours Post First Dose at Day 1 (4 Hours Post First Dose), and 2, 4, 8, 11, 15, 18, 22 and 25: DB Treatment Phase
Description: CGI-SS-R is revised version of the CGI-S. The CGI-SS-R summarizes the clinician's overall impression of severity of suicidality on a 7-point scale from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal participants), based on the totality of information available to the clinician. A higher score indicates a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1, predose), Days 1 (4 hours postdose), 2, 4, 8, 11, 15, 18, 22 and 25
Population: as for outcome 4
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 1: 4 hours postdose: number analyzed (Participants) | 112 | 112
  Change at Day 1: 4 hours postdose | -1.0 [-4 to 1] | -1.0 [-6 to 1]
  Change at Day 2: number analyzed (Participants) | 111 | 108
  Change at Day 2 | -1.0 [-5 to 2] | -1.0 [-6 to 2]
  Change at Day 4: number analyzed (Participants) | 111 | 107
  Change at Day 4 | -2.0 [-5 to 2] | -2.0 [-6 to 1]
  Change at Day 8: number analyzed (Participants) | 105 | 99
  Change at Day 8 | -2.0 [-5 to 2] | -2.0 [-5 to 2]
  Change at Day 11: number analyzed (Participants) | 99 | 95
  Change at Day 11 | -2.0 [-6 to 2] | -3.0 [-6 to 1]
  Change at Day 15: number analyzed (Participants) | 99 | 91
  Change at Day 15 | -3.0 [-5 to 2] | -3.0 [-6 to 0]
  Change at Day 18: number analyzed (Participants) | 90 | 84
  Change at Day 18 | -3.0 [-6 to 1] | -3.0 [-5 to 0]
  Change at Day 22: number analyzed (Participants) | 95 | 90
  Change at Day 22 | -3.0 [-5 to 3] | -3.0 [-5 to 0]
  Change at Day 25: number analyzed (Participants) | 88 | 85
  Change at Day 25 | -3.0 [-6 to 4] | -3.0 [-6 to 0]

6. Secondary Outcome: Number of Participants Who Achieved Resolution of Suicidality (CGI-SS-R Score of 0 or 1): DB Treatment Phase
Description: CGI-SS-R is revised version of the CGI-S. The CGI-SS-R summarizes the clinician's overall impression of severity of suicidality on a 7-point scale from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal participants), based on the totality of information available to the clinician. Higher score indicates a more severe condition. A participant was considered to have achieved resolution of suicidality at a given time point if the CGI-SS-R score was 0 (normal, not at all suicidal) or 1 (questionably suicidal). Participants who did not met such criterion or discontinued prior to the time point for any reason were not considered to have resolution of suicidality.
Time Frame: Days 1 (4 hours postdose), 2, 4, 8, 11, 15, 18, 22 and 25
Population: Analysis was performed on full efficacy analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
Participants
  Day 1: 4 hours postdose | 20 | 38
  Day 2 | 35 | 36
  Day 4 | 51 | 52
  Day 8 | 54 | 53
  Day 11 | 58 | 62
  Day 15 | 58 | 65
  Day 18 | 59 | 62
  Day 22 | 65 | 68
  Day 25 | 66 | 69

7. Secondary Outcome: Change From Baseline in Clinical Global Impression of Imminent Suicide Risk (CGI-SR-I) at Days 1, 2, 4, 8, 11, 15, 18, 22 and 25: DB Treatment Phase
Description: The CGI-SR-I is a scale summarizing the clinician's best assessment of the likelihood that the participant will attempt suicide in the next 7 days. The CGI-SR-I rating is scored on a 7-point scale: where' 0 (no imminent suicide risk); 1 (minimal imminent suicide risk), 2 (mild imminent suicide risk), 3 (moderate imminent suicide risk), 4 (marked imminent suicide risk), 5 (severely imminent suicide risk), 6 (extreme imminent suicide risk). Higher score indicates a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1, predose), Days 1 (4 hours postdose), 2, 4, 8, 11, 15, 18, 22 and 25
Population: Analysis was performed on full efficacy analysis set. Here, 'n' (number analyzed) signifies the number of participants analyzed at each specified time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 1: 4 hours postdose: number analyzed (Participants) | 112 | 112
  Change at Day 1: 4 hours postdose | 0.0 [-4 to 2] | -1.0 [-6 to 3]
  Change at Day 2: number analyzed (Participants) | 111 | 108
  Change at Day 2 | -1.0 [-4 to 2] | -1.0 [-6 to 2]
  Change at Day 4: number analyzed (Participants) | 111 | 107
  Change at Day 4 | -2.0 [-5 to 2] | -2.0 [-6 to 1]
  Change at Day 8: number analyzed (Participants) | 105 | 98
  Change at Day 8 | -2.0 [-5 to 2] | -2.0 [-5 to 2]
  Change at Day 11: number analyzed (Participants) | 99 | 95
  Change at Day 11 | -2.0 [-5 to 1] | -2.0 [-6 to 2]
  Change at Day 15: number analyzed (Participants) | 99 | 95
  Change at Day 15 | -3.0 [-5 to 2] | -2.0 [-6 to 1]
  Change at Day 18: number analyzed (Participants) | 90 | 84
  Change at Day 18 | -3.0 [-5 to 2] | -3.0 [-5 to 1]
  Change at Day 22: number analyzed (Participants) | 95 | 90
  Change at Day 22 | -3.0 [-5 to 2] | -3.0 [-5 to 0]
  Change at Day 25: number analyzed (Participants) | 88 | 85
  Change at Day 25 | -3.0 [-5 to 2] | -3.0 [-6 to 1]

8. Secondary Outcome: Change From Baseline in Beck Hopelessness Scale (BHS) Total Score at Days 8 and 25 in DB Treatment Phase
Description: BHS is a self-reported measure to assess one's level of negative expectations or pessimism regarding future. It consists of 20 true-false items that examine respondent's attitude over past week by either endorsing a pessimistic statement or denying an optimistic statement; 9 are keyed false and 11 are keyed true. For every statement, each response was assigned score of 0 or 1. Total BHS score is sum of item responses, ranged from 0-20, where higher score represented higher level of hopelessness.
Time Frame: Baseline, Days 8 and 25
Population: Analysis was performed on full efficacy analysis set. Here, 'n' (number analyzed) signifies number of participants analyzed for each specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 8: number analyzed (Participants) | 108 | 104
  Change at Day 8 | -6.3 (6.31) | -6.1 (6.17)
  Change at Day 25: number analyzed (Participants) | 96 | 91
  Change at Day 25 | -7.0 (6.47) | -8.0 (6.31)

9. Secondary Outcome: Change From Baseline in European Quality of Life Group, 5-Dimension, 5-Level (EQ-5D-5L) Sum Score at Days 2, 11 and 25 of the DB Treatment Phase
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). EQ-5D-5L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (no problem, slight, moderate, severe and extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate Health Status Index (HSI). HSI ranges from 0 (dead) to 1.00 (full health). EQ-VAS self-rating records respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst imaginable health)-100 (best imaginable health). Sum score ranges from 0 -100. Sum score=(sum of the scores from the 5 dimensions minus 5)*5. Higher score indicates worse health state. Negative change in score indicates improvement.
Time Frame: Baseline, Days 2, 11 and 25
Population: Analysis was performed on full efficacy analysis set. Here, 'n' (number analyzed) signifies the number of participants analyzed for each specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 2: number analyzed (Participants) | 111 | 107
  Change at Day 2 | -9.0 (12.30) | -11.8 (14.45)
  Change at Day 11: number analyzed (Participants) | 103 | 103
  Change at Day 11 | -15.1 (16.32) | -15.0 (15.51)
  Change at Day 25: number analyzed (Participants) | 95 | 92
  Change at Day 25 | -15.3 (15.78) | -18.8 (16.96)

10. Secondary Outcome: Change From Baseline in European Quality of Life Group, Visual Analogue Scale (EQ-VAS) Score at Days 2, 11 and 25 of the DB Treatment Phase
Description: EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. The EQ VAS self-rating records the respondent's own assessment of his or her overall health status at the time of completion, on a scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine). Positive change in score indicates improvement.
Time Frame: Baseline, Days 2, 11 and 25
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 2: number analyzed (Participants) | 111 | 107
  Change at Day 2 | 9.7 (15.57) | 13.4 (22.58)
  Change at Day 11: number analyzed (Participants) | 103 | 103
  Change at Day 11 | 17.6 (24.87) | 21.4 (26.95)
  Change at Day 25: number analyzed (Participants) | 95 | 92
  Change at Day 25 | 18.6 (25.39) | 27.0 (27.54)

11. Secondary Outcome: Change From Baseline in EQ-5D-5L Health Status Index at Days 2, 11 and 25 of the DB Treatment Phase
Description: EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a HSI. HSI ranges from 0 (dead) to 1.00 (full health). Positive change in score indicates improvement.
Time Frame: Baseline, Days 2, 11 and 25
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 2: number analyzed (Participants) | 111 | 107
  Change at Day 2 | 0.129 (0.1732) | 0.160 (0.1872)
  Change at Day 11: number analyzed (Participants) | 103 | 103
  Change at Day 11 | 0.194 (0.2173) | 0.202 (0.2051)
  Change at Day 25: number analyzed (Participants) | 95 | 92
  Change at Day 25 | 0.194 (0.2149) | 0.235 (0.2228)

12. Secondary Outcome: Change From Baseline in Quality of Life in Depression Scale (QLDS) Total Score at Days 2, 11 and 25 of the DB Treatment Phase
Description: The QLDS is a disease-specific patient-reported outcome designed to assess health-related quality of life in patients with MDD, it captures the impact of depression and its treatment from the participant's perspective. The instrument has a recall period of "at the moment" and contains 34 items with "true"/"not true" response options. The total score range is from 0 (good quality of life) to 34 (very poor quality of life). A higher score indicates a more severe condition. Negative change indicates improvement.
Time Frame: Baseline, Days 2, 11 and 25
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 2: number analyzed (Participants) | 111 | 107
  Change at Day 2 | -2.5 (3.93) | -3.5 (4.93)
  Change at Day 11: number analyzed (Participants) | 103 | 103
  Change at Day 11 | -5.2 (5.55) | -5.1 (6.16)
  Change at Day 25: number analyzed (Participants) | 95 | 92
  Change at Day 25 | -5.5 (6.03) | -6.3 (6.26)

13. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM-9) Domain Score at Days 15 and 25: DB Treatment Phase
Description: The TSQM-9 is a 9-item generic patient-reported outcome instrument to assess participants' satisfaction with medication. It covers domains of effectiveness, convenience, and global satisfaction. The TSQM-9 domain scores were calculated as recommended by the instrument authors. (i) Effectiveness = [(item 1 + item 2 + item 3) - 3]/18*100, (ii) Convenience = [(item 4 + item 5 + item 6) - 3]/18*100 and (iii) Global satisfaction = [(item 7 + item 8 + item 9) - 3]/14*100. Each domain score can be calculated only if all the three items considered in the calculation of that score are not missing. The TSQM-9 domain score ranges from 0 to 100, with higher scores representing higher satisfaction.
Time Frame: Days 15 and 25
Population: Analysis was performed on full efficacy analysis. Here, 'n' (number analyzed) signifies the number of participants analyzed for each specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Effectiveness: Day 15: number analyzed (Participants) | 97 | 101
  Effectiveness: Day 15 | 55.3 (27.93) | 63.5 (26.05)
  Effectiveness: Day 25: number analyzed (Participants) | 113 | 90
  Effectiveness: Day 25 | 54.8 (28.84) | 68.8 (25.41)
  Convenience: Day 15 | 77.2 (16.73) | 71.3 (18.38)
  Convenience: Day 25: number analyzed (Participants) | 113 | 90
  Convenience: Day 25 | 76.9 (17.92) | 77.0 (18.66)
  Global Satisfaction: Day 15 | 59.7 (27.12) | 63.6 (27.69)
  Global Satisfaction: Day 25: number analyzed (Participants) | 113 | 90
  Global Satisfaction: Day 25 | 56.8 (28.31) | 71.5 (24.85)

14. Secondary Outcome: Change From Baseline in Suicide Ideation and Behavior Assessment Tool (SIBAT) Module 5 (My Risk) Question 3 (Participant-Reported Frequency of Suicidal Thinking) Score at Days 1, 2, 4, 8, 11, 15, 18, 22 and 25: DB Treatment Phase
Description: SIBAT is an assessment tool that captures suicidal ideation, behavior, and risk. It permits assessment of change in suicidal ideation and behavior and documents clinician assessment of severity of suicidality and suicide risk. SIBAT is organized into 8 modules divided into 2 major divisions: patient-reported section (Modules 1-5) and clinician-rated section (Modules 6-8). Patient-reported section has modules of demographics and suicide history, risk/protective factors, suicidal thinking, suicide behavior, and suicide risk. Question 3 from Module 5 asks participants to describe their thinking about suicide right now from 5 response options ranging from 0 (I have no suicidal thoughts) to 4 (I have suicidal thoughts all of time).
Time Frame: Baseline, Days 1 (4h postdose), 2, 4, 8, 11, 15, 18, 22 and 25
Population: as for outcome 9
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 1: 4 hours postdose: number analyzed (Participants) | 111 | 109
  Change at Day 1: 4 hours postdose | -1.0 [-3 to 1] | -1.0 [-4 to 2]
  Change at Day 2: number analyzed (Participants) | 110 | 106
  Change at Day 2 | -1.0 [-4 to 1] | -1.0 [-4 to 2]
  Change at Day 4: number analyzed (Participants) | 109 | 107
  Change at Day 4 | -1.0 [-4 to 1] | -1.0 [-4 to 4]
  Change at Day 8: number analyzed (Participants) | 105 | 98
  Change at Day 8 | -2.0 [-4 to 1] | -2.0 [-4 to 4]
  Change at Day 11: number analyzed (Participants) | 97 | 96
  Change at Day 11 | -2.0 [-4 to 1] | -2.0 [-4 to 4]
  Change at Day 15: number analyzed (Participants) | 96 | 92
  Change at Day 15 | -2.0 [-4 to 0] | -2.0 [-4 to 1]
  Change at Day 18: number analyzed (Participants) | 89 | 83
  Change at Day 18 | -2.0 [-4 to 2] | -2.0 [-4 to 3]
  Change at Day 22: number analyzed (Participants) | 96 | 90
  Change at Day 22 | -2.0 [-4 to 1] | -2.0 [-4 to 3]
  Change at Day 25: number analyzed (Participants) | 88 | 84
  Change at Day 25 | -2.0 [-4 to 1] | -2.0 [-4 to 4]

15. Secondary Outcome: Change From Baseline in Suicide Ideation and Behavior Assessment Tool (SIBAT) Module 7 (Clinician-rated Frequency of Suicidal Thinking [FoST]) Score at Days 1, 2, 4, 8, 11, 15, 18, 22 and 25: DB Treatment Phase
Description: SIBAT is assessment tool that captures suicidal ideation, behavior, and risk. It permits assessment of change in suicidal ideation and behavior and documents clinician assessment of severity of suicidality and suicide risk. SIBAT has 8 modules divided into 2 major divisions: patient-reported section (Modules 1-5) and clinician-rated section (Modules 6-8). Clinician-rated section has modules for semi-structured interview, clinical global impressions of current severity of suicidality and imminent suicide risk, clinical global impression of long-term suicide risk, and clinical judgment of optimal suicide management. The score anchor point as in participant report frequency of suicidal thinking that is, response options from never to all the time. Module 7-FoST score ranges from 0-5; higher score indicates more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline, Days 1 (4 hours postdose), 2, 4, 8, 11, 15, 18, 22 and 25
Population: as for outcome 9
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
units on a scale
  Change at Day 1: 4 hours postdose: number analyzed (Participants) | 112 | 112
  Change at Day 1: 4 hours postdose | -1.0 [-4 to 2] | -1.0 [-5 to 1]
  Change at Day 2: number analyzed (Participants) | 111 | 108
  Change at Day 2 | -1.0 [-5 to 1] | -1.0 [-5 to 1]
  Change at Day 4: number analyzed (Participants) | 111 | 107
  Change at Day 4 | -2.0 [-5 to 1] | -2.0 [-5 to 1]
  Change at Day 8: number analyzed (Participants) | 105 | 99
  Change at Day 8 | -2.0 [-4 to 1] | -2.0 [-5 to 1]
  Change at Day 11: number analyzed (Participants) | 99 | 95
  Change at Day 11 | -2.0 [-5 to 2] | -2.0 [-5 to 1]
  Change at Day 15: number analyzed (Participants) | 99 | 91
  Change at Day 15 | -2.0 [-5 to 2] | -3.0 [-5 to 0]
  Change at Day 18: number analyzed (Participants) | 90 | 84
  Change at Day 18 | -2.0 [-5 to 1] | -3.0 [-5 to 1]
  Change at Day 22: number analyzed (Participants) | 95 | 90
  Change at Day 22 | -2.0 [-5 to 2] | -3.0 [-5 to 2]
  Change at Day 25: number analyzed (Participants) | 88 | 85
  Change at Day 25 | -2.0 [-5 to 4] | -3.0 [-5 to 2]

16. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): DB Treatment Phase
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. A TEAE is categorized as related if assessed by the investigator as possibly, probably, or very likely related to study agent.
Time Frame: Up to Day 25
Population: Safety analysis set (SAS) included all randomized participants who received at least 1 dose of study drug in the DB treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
Participants | 87 | 104

17. Secondary Outcome: Number of Participants With Treatment Emergent Abnormal Laboratory Values: DB Treatment Phase
Description: Low/high abnormal values are: Alanine aminotransferase (ALT)-high=200 Units per liter(U/L); ALP-high=250U/L; aspartate aminotransferase(AST)-high=250U/L; gamma glutamyl transferase(GGT)=300U/L; Albumin (low=24g/L,high=60 g/L); Bicarbonate(low=15.1, high=34.9mmol/L); Bilirubin(high=51.3micromol/L); calcium(low=1.5,high=3mmol/L);Chloride(low=94,high=112mmol/L); CK(High=990U/L); Creatinine (High=265.2micromol/L); Eosinophils(High=10%); Erythrocytes(low=3.0*1012/L,high=6.4*1012/L); Glucose(low=2.2,high=16.7mmol/L); Hemoglobin(low=80g/L,high=190g/L);Hematocrit(low=0.28, high=0.55 fraction); LD(high=500U/L); Leukocytes(low=2.5*109/L,high=15.5*109/L); Lymphocytes(low=10%,high=60%); Monocytes(high=20%); Neutrophils(low=30%,high=90%); Phosphate(low=0.7 mmol/L,high=2.6mmol/L); Platelet count(low=100*109/L,high=600*109/L]; Potassium(low=3.0mmol/L,high=5.8 mmol/L]; Protein(low=50 g/L); Sodium(low=125 mmol/L,high=155 mmol/L); Urate(low=89.2 micromol/L,high=594.8micromol/L); Urine(high=8.0 pH).
Time Frame: Up to Day 25
Population: SAS: all randomized participants who received at least 1 dose of study drug in DB phase. 'N'(number of participants analyzed) signifies number of participants analyzed for this OM. 'n' (number analyzed) signifies number of participants analyzed for each specified category. mmol/L=millimoles per liter; g/L=gram per liter; ULN=upper limit of normal
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 101 | 101
Participants
  ALT: ALT>3*ULN: number analyzed (Participants) | 92 | 97
  ALT: ALT>3*ULN | 2 | 2
  ALT: Abnormal High: number analyzed (Participants) | 92 | 97
  ALT: Abnormal High | 0 | 0
  Albumin: Abnormal High | 0 | 0
  Albumin: Abnormal Low | 0 | 0
  Alkaline phosphatase (ALP): Abnormal High: number analyzed (Participants) | 99 | 99
  Alkaline phosphatase (ALP): Abnormal High | 0 | 0
  AST: AST>3*ULN: number analyzed (Participants) | 90 | 97
  AST: AST>3*ULN | 0 | 0
  AST: Abnormal High: number analyzed (Participants) | 90 | 97
  AST: Abnormal High | 0 | 0
  Bicarbonate: Abnormal High: number analyzed (Participants) | 91 | 96
  Bicarbonate: Abnormal High | 0 | 0
  Bicarbonate: Abnormal Low: number analyzed (Participants) | 91 | 96
  Bicarbonate: Abnormal Low | 0 | 0
  Bilirubin: Abnormal High: number analyzed (Participants) | 92 | 97
  Bilirubin: Abnormal High | 0 | 0
  Calcium: Abnormal High: number analyzed (Participants) | 99 | 99
  Calcium: Abnormal High | 0 | 0
  Calcium: Abnormal Low: number analyzed (Participants) | 99 | 99
  Calcium: Abnormal Low | 0 | 0
  Chloride: Abnormal High: number analyzed (Participants) | 99 | 99
  Chloride: Abnormal High | 0 | 0
  Chloride: Abnormal Low: number analyzed (Participants) | 99 | 99
  Chloride: Abnormal Low | 0 | 0
  Creatine Kinase (CK): Abnormal High: number analyzed (Participants) | 92 | 97
  Creatine Kinase (CK): Abnormal High | 0 | 0
  Creatinine: Abnormal High: number analyzed (Participants) | 99 | 99
  Creatinine: Abnormal High | 0 | 0
  GGT: Abnormal High: number analyzed (Participants) | 99 | 99
  GGT: Abnormal High | 3 | 1
  Glucose: Abnormal High: number analyzed (Participants) | 92 | 97
  Glucose: Abnormal High | 0 | 1
  Glucose: Abnormal Low: number analyzed (Participants) | 92 | 97
  Glucose: Abnormal Low | 0 | 0
  ALT>3*ULN or AST>3*ULN and BILI>2*ULN: number analyzed (Participants) | 92 | 97
  ALT>3*ULN or AST>3*ULN and BILI>2*ULN | 0 | 0
  Lactate Dehydrogenase (LD): Abnormal High: number analyzed (Participants) | 86 | 89
  Lactate Dehydrogenase (LD): Abnormal High | 0 | 0
  Phosphate: Abnormal High | 0 | 0
  Phosphate: Abnormal Low | 0 | 1
  Potassium: Abnormal High: number analyzed (Participants) | 99 | 99
  Potassium: Abnormal High | 1 | 0
  Potassium: Abnormal Low: number analyzed (Participants) | 99 | 99
  Potassium: Abnormal Low | 0 | 0
  Protein: Abnormal Low: number analyzed (Participants) | 99 | 99
  Protein: Abnormal Low | 0 | 0
  Sodium: Abnormal High: number analyzed (Participants) | 99 | 99
  Sodium: Abnormal High | 0 | 0
  Sodium: Abnormal Low: number analyzed (Participants) | 99 | 99
  Sodium: Abnormal Low | 0 | 0
  Urate: Abnormal High: number analyzed (Participants) | 99 | 99
  Urate: Abnormal High | 0 | 0
  Urate: Abnormal Low: number analyzed (Participants) | 99 | 99
  Urate: Abnormal Low | 0 | 0
  Basophils: Abnormal High: number analyzed (Participants) | 87 | 94
  Basophils: Abnormal High | 0 | 0
  Eosinophils: Abnormal High: number analyzed (Participants) | 87 | 94
  Eosinophils: Abnormal High | 0 | 0
  Erythrocytes: Abnormal High: number analyzed (Participants) | 84 | 94
  Erythrocytes: Abnormal High | 0 | 1
  Erythrocytes: Abnormal Low: number analyzed (Participants) | 87 | 94
  Erythrocytes: Abnormal Low | 0 | 0
  Hematocrit: Abnormal High: number analyzed (Participants) | 86 | 92
  Hematocrit: Abnormal High | 0 | 2
  Hematocrit: Abnormal Low: number analyzed (Participants) | 86 | 92
  Hematocrit: Abnormal Low | 0 | 0
  Hemoglobin (Hb): Abnormal High: number analyzed (Participants) | 87 | 94
  Hemoglobin (Hb): Abnormal High | 0 | 1
  Hemoglobin: Abnormal Low: number analyzed (Participants) | 87 | 94
  Hemoglobin: Abnormal Low | 0 | 0
  Leukocytes: Abnormal High: number analyzed (Participants) | 87 | 94
  Leukocytes: Abnormal High | 1 | 0
  Leukocytes: Abnormal Low: number analyzed (Participants) | 87 | 94
  Leukocytes: Abnormal Low | 0 | 0
  Lymphocytes: Abnormal High: number analyzed (Participants) | 87 | 94
  Lymphocytes: Abnormal High | 0 | 0
  Lymphocytes: Abnormal Low: number analyzed (Participants) | 87 | 94
  Lymphocytes: Abnormal Low | 2 | 1
  Monocytes: Abnormal High: number analyzed (Participants) | 87 | 94
  Monocytes: Abnormal High | 0 | 0
  Neutrophils: Abnormal High: number analyzed (Participants) | 87 | 94
  Neutrophils: Abnormal High | 0 | 0
  Neutrophils: Abnormal Low: number analyzed (Participants) | 87 | 94
  Neutrophils: Abnormal Low | 0 | 1
  Platelets: Abnormal High: number analyzed (Participants) | 87 | 94
  Platelets: Abnormal High | 0 | 0
  Platelets: Abnormal Low: number analyzed (Participants) | 87 | 94
  Platelets: Abnormal Low | 0 | 1
  Urine pH: Abnormal High: number analyzed (Participants) | 96 | 97
  Urine pH: Abnormal High | 0 | 0

18. Secondary Outcome: Number of Participants With Abnormal Nasal Examinations at Day 25: DB Treatment Phase
Description: Number of participants with abnormal nasal examination were reported. Nasal examination of visual inspection of the epistaxis, nasal crusts, nasal discharge, and nasal erythema was performed.
Time Frame: At Day 25
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug in the DB treatment phase. Here, 'n' (number analyzed) signifies number of participants analyzed for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
Participants
  Epistaxis: Mild: number analyzed (Participants) | 105 | 104
  Epistaxis: Mild | 1 | 1
  Epistaxis: Moderate: number analyzed (Participants) | 105 | 104
  Epistaxis: Moderate | 0 | 0
  Epistaxis: Severe: number analyzed (Participants) | 105 | 104
  Epistaxis: Severe | 0 | 0
  Nasal Crusts: Mild: number analyzed (Participants) | 105 | 104
  Nasal Crusts: Mild | 0 | 1
  Nasal Crusts: Moderate: number analyzed (Participants) | 105 | 104
  Nasal Crusts: Moderate | 0 | 0
  Nasal Crusts: Severe: number analyzed (Participants) | 105 | 104
  Nasal Crusts: Severe | 0 | 0
  Nasal Discharge: Mild: number analyzed (Participants) | 105 | 104
  Nasal Discharge: Mild | 0 | 1
  Nasal Discharge: Moderate: number analyzed (Participants) | 105 | 104
  Nasal Discharge: Moderate | 0 | 0
  Nasal Discharge: Severe: number analyzed (Participants) | 105 | 104
  Nasal Discharge: Severe | 0 | 0
  Nasal Erythema: Mild: number analyzed (Participants) | 105 | 104
  Nasal Erythema: Mild | 1 | 4
  Nasal Erythema: Moderate: number analyzed (Participants) | 105 | 104
  Nasal Erythema: Moderate | 1 | 0
  Nasal Erythema: Severe: number analyzed (Participants) | 105 | 104
  Nasal Erythema: Severe | 0 | 0

19. Secondary Outcome: Number of Participants With Treatment Emergent Abnormal Electrocardiogram (ECG) Values at Any Time: DB Treatment Phase
Description: Number of participants with treatment emergent abnormal ECG values for variables including heart rate (abnormally low refers to less than or equal to [<=] 50 beats per minute [bpm] , abnormally high refers greater than or equal to [>=] 100 bpm), pulse rate (PR) interval (abnormally high refers to >= 210 milliseconds [msec]), QRS interval (abnormally Low refers to <= 50, abnormally high refers to >= 120 msec) and QT interval (abnormally low refers to <= 200, abnormally high >= 500 msec) were reported.
Time Frame: Up to Day 25
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug in the DB treatment phase. Here 'N' (number of participants analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 112
Participants
  Heart Rate <= 50 bpm | 9 | 2
  Heart Rate >= 100 bpm | 3 | 2
  PR Duration >= 210 msec | 2 | 2
  QRS Duration <= 50 msec | 0 | 0
  QRS Duration >= 120 msec | 1 | 0
  QT Duration <= 200 msec | 0 | 0
  QT Duration >= 500 msec | 0 | 0

20. Secondary Outcome: Number of Participants With Abnormal Arterial Oxygen Saturation (SpO2) Levels (Less Than [<] 93%) as Assessed by Pulse Oximetry at Any Time: DB Treatment Phase
Description: Pulse oximetry was used to measure arterial SpO2 levels. On each dosing day, the device was attached to the finger, toe, or ear, and SpO2 was monitored and documented. If oxygen saturation levels were less than (<) 93% at any time during the 1.5 hours postdose interval, pulse oximetry was recorded every 5 minutes until levels return to >= 93% or until the participant is referred for appropriate medical care, if clinically indicated. Participants with at least 2 consecutive postdose oxygen saturation below 93% during the DB treatment phase were reported.
Time Frame: Up to Day 25
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug in the DB treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
Participants | 2 | 3

21. Secondary Outcome: Number of Participants With Treatment Emergent Vital Signs Abnormalities: DB Treatment Phase
Description: Number of participants with treatment emergent vital signs abnormalities (pulse rate in bpm [abnormally low = a decrease from baseline of >= 15 to a value <= 50; abnormally high = an increase from baseline of >=15 to a value >=100] , systolic blood pressure [SBP] in mmHg [abnormally low = a decrease from baseline of >= 20 to a value <= 90; abnormally high = an increase from baseline of >= 20 to a value >= 180], and diastolic blood pressure [DBP] in mmHg [abnormally low= a decrease from baseline of >=15 to a value <= 50; abnormally high = an increase from baseline of >= 15 to a value >= 105) were reported.
Time Frame: Up to Day 25
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
Participants
  Pulse rate (bpm): Decrease of >=15 to <=50 | 2 | 1
  Pulse rate (bpm): Increase of >=15 to >=100 | 11 | 12
  SBP: Decrease of >=20 to <=90 | 5 | 2
  SBP (mmHg): Increase of >=20 to >=180 | 2 | 3
  DBP (mmHg): Decrease of >=15 to <=50 | 4 | 4
  DBP (mmHg): Increase of >=15 to >=105 | 3 | 6

22. Secondary Outcome: Number of Sedated Participants as Assessed by Modified Observer's Assessment of Alertness/Sedation (MOAA/S) Score at Any Time: DB Treatment Phase
Description: MOAA/S was used to measure treatment-emergent sedation with correlation to levels of sedation defined by the American society of anesthesiologists (ASA) continuum. The MOAA/S scores range from 0 to 5 where,0 = no response to painful stimulus; ASA continuum = general anesthesia, 1 = responds to trapezius squeeze; ASA continuum = deep sedation, 2 = purposeful response to mild prodding or mild shaking; ASA continuum = moderate sedation, 3 = responds after name called loudly or repeatedly; ASA continuum = moderate sedation, 4 = lethargic response to name spoken in normal tone; ASA continuum = moderate sedation and 5 = readily responds to name spoken in normal tone (awake); ASA continuum = minimal sedation.
Time Frame: Up to Day 25
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
Participants
  Score <=2: Yes | 0 | 4
  Score <=3: Yes | 3 | 21
  Score <=4: Yes | 20 | 65

23. Secondary Outcome: Number of Participants With an Increase in Clinician-administered Dissociative States Scale (CADSS) Total Score Over Time: DB Treatment Phase
Description: The CADSS used to measure present-state dissociative symptoms, and to assess treatment-emergent dissociative symptoms. It comprises 23 subjective items divided into 3 components: depersonalization (with score range from 0 to 28), derealization (with score range from 0 to 52), and amnesia (with score range from 0 to 8). Participants responses are coded on a 5-point scale (0 = "Not at all", 1 = "Mild", 2 = "Moderate", 3 = 'Severe" and 4 = "Extreme"). The total score is sum of the 23 items and range from 0 to 92, where 0 (best) and 92 (worst). A higher score indicates a more severe condition. Number of participants with an increase in CADSS total score (increase based on maximum CADSS total score change from predose of > 0) was reported.
Time Frame: Days 1, 4, 8, 11, 15, 18, 22 and 25
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug in the DB treatment phase. Here, 'n' (number analyzed) signifies the number of participants analyzed for each specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
Number analyzed (Participants) | 113 | 114
Participants
  Day 1: number analyzed (Participants) | 111 | 113
  Day 1 | 28 | 106
  Day 4: number analyzed (Participants) | 105 | 104
  Day 4 | 21 | 86
  Day 8: number analyzed (Participants) | 106 | 98
  Day 8 | 16 | 75
  Day 11: number analyzed (Participants) | 96 | 90
  Day 11 | 8 | 68
  Day 15: number analyzed (Participants) | 96 | 91
  Day 15 | 11 | 68
  Day 18: number analyzed (Participants) | 88 | 80
  Day 18 | 8 | 53
  Day 22: number analyzed (Participants) | 93 | 89
  Day 22 | 7 | 58
  Day 25: number analyzed (Participants) | 88 | 85
  Day 25 | 4 | 56

ADVERSE EVENTS:
Time Frame: Up to Day 25
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug in the double-blind treatment phase.
Arm/Group | Placebo + Standard of Care (SOC) | Esketamine 84 mg + SOC
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/114
Serious Adverse Events (participants affected / at risk) | 6/113 | 5/114
Other Adverse Events (participants affected / at risk) | 74/113 | 98/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Standard of Care (SOC) (N=113) | Esketamine 84 mg + SOC (N=114)
Arrhythmia (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Depersonalisation/Derealisation Disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 2 | 1
Suicide Attempt (Psychiatric disorders) | 3 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Standard of Care (SOC) (N=113) | Esketamine 84 mg + SOC (N=114)
Vertigo (Ear and labyrinth disorders) | 0 | 7
Diplopia (Eye disorders) | 0 | 6
Vision Blurred (Eye disorders) | 6 | 17
Constipation (Gastrointestinal disorders) | 9 | 7
Dry Mouth (Gastrointestinal disorders) | 5 | 8
Hypoaesthesia Oral (Gastrointestinal disorders) | 2 | 7
Nausea (Gastrointestinal disorders) | 16 | 38
Paraesthesia Oral (Gastrointestinal disorders) | 3 | 14
Vomiting (Gastrointestinal disorders) | 5 | 18
Feeling Drunk (General disorders) | 1 | 6
Blood Pressure Increased (Investigations) | 3 | 7
Dizziness (Nervous system disorders) | 21 | 47
Dizziness Postural (Nervous system disorders) | 1 | 9
Dysgeusia (Nervous system disorders) | 18 | 29
Headache (Nervous system disorders) | 26 | 25
Hypoaesthesia (Nervous system disorders) | 1 | 12
Paraesthesia (Nervous system disorders) | 7 | 23
Sedation (Nervous system disorders) | 3 | 16
Somnolence (Nervous system disorders) | 12 | 26
Anxiety (Psychiatric disorders) | 7 | 17
Depersonalisation/Derealisation Disorder (Psychiatric disorders) | 0 | 9
Dissociation (Psychiatric disorders) | 9 | 44
Euphoric Mood (Psychiatric disorders) | 1 | 13
Insomnia (Psychiatric disorders) | 11 | 9
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 6

LIMITATIONS AND CAVEATS:
Esketamine's known characteristic effects such as dissociative symptoms, sedation, and elevation of blood pressure may have impact on blinding, to minimize this bias, protocol specified that different raters perform efficacy and safety assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT03097133/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT03097133/SAP_001.pdf